CLINICAL TRIAL: NCT05260411
Title: A Phase 3 Clinical Study Evaluating the Efficacy and Safety of AK102 Q6W in Patients With Primary Hypercholesterolemia and Mixed Hyperlipidemia
Brief Title: A Study to Evaluate the Efficacy and Safety of AK102 Q6W in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK102-302
Record Dates: First submitted 2022-02-09; First posted 2022-03-02 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AK102 regimen 1 (Experimental)
  Interventions: Biological: AK102
- AK102 regimen 2 (Experimental)
  Interventions: Biological: AK102
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AK102 — Administered AK102 450 mg by subcutaneous injection every 6 weeks Drug: Statins and/or Ezetimibe lipid-lowering therapies
  Arms: AK102 regimen 1
Biological: AK102 — Administered AK102 600 mg by subcutaneous injection every 6 weeks Drug: Statins and/or Ezetimibe lipid-lowering therapies
  Arms: AK102 regimen 2
Drug: Placebo — Administered placebo by subcutaneous injection every 6 weeks Drug: Statins and/or Ezetimibe lipid-lowering therapies
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase # clinical study evaluating the efficacy and safety of AK102 Q6W in patients with primary hypercholesterolemia and mixed hyperlipidemia.

DETAILED DESCRIPTION:
This is a Phase 3 clinical study to evaluate the efficacy and safety of AK102 Q6W, a monoclonal antibody against proprotein convertase subtilisin/kexin type 9 (PCSK9), in subjects with primary hypercholesterolemia and mixed hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject understand and voluntarily sign the written Inform Consent Form (ICF).
2. Male or female ≥ 18 to ≤ 80 years of age.
3. The fasting serum LDL-C level of subjects did not meet the treatment goal after at least 4 weeks of stable lipid-lowering background treatment.
4. TG ≤ 4.5 mmol/L (400 mg/dl)

Exclusion Criteria:

1. Known homozygous familial hypercholesterolemia.
2. Received PCSK9 inhibitors within 6 months before randomization.
3. Known sensitivity to PCSK9 inhibitors and any substances to be administered.
4. Severe renal dysfunction.
5. Previously received organ transplantation.
6. Uncontrolled hypothyroidism or hyperthyroidism.
7. Uncontrolled hypertension.
8. Known hyperlipidemia secondary to comorbidity, including nephrotic syndrome, cholestatic liver failure, etc.
9. History of malignancy of any organ system within the past 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 246 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline of serum LDL-C level | At week 12

SECONDARY OUTCOMES:
Percentage change from baseline of serum LDL-C, TC, HDL-C, TG, ApoB, ApoA-I, non HDL-C and Lp(a) levels | Week 0-24
The incidence and severity of adverse events (AE) | Week 0-24
Evaluate the changes of AK102 PK parameters(t1/2) | Week 0-24
Evaluate the changes of AK102 PK parameters(AUC） | Week 0-24
Evaluate the changes of AK102 PK parameters(Vd) | Week 0-24
Evaluate the changes of AK102 PK parameters(Tmax) | Week 0-24
Evaluate the changes of free PCSK9 concentration | Week 0-24
Evaluate the changes of AK102 PK parameters(Cmax) | Week 0-24
Evaluate the changes of AK102 PK parameters(CL) | Week 0-24
Evaluate the changes of AK102 PK parameters(MRT) | Week 0-24
The number and percentage of anti AK102 antibody (ADA)positive subjects | Week 0-24
The number and percentage of anti AK102 neutralizing antibody (NAB) positive subjects | Week 0-24
the time of ADA positive | Week 0-24
the time of nab positive | Week 0-24

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhongshan Hospital, Fudan Hospital, Shanghai